CLINICAL TRIAL: NCT07014384
Title: A Randomized, Sham-controlled Study of Cerebellar Transcranial Direct Current Stimulation (tDCS) and Its Effects on the Neurophysiological Properties of the Sensorimotor Network and Motor Symptom Severity in Patients With Isolated Cervical Dystonia (CD)
Brief Title: Cerebellar Transcranial Direct Current Stimulation (tDCS) in Patients With Isolated Cervical Dystonia (CD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Simone Zittel, Dr. med., Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Cereb_tDCS_in_CD
Record Dates: First submitted 2025-05-19; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Isolated Cervical Dystonia
Keywords: Isolated Cervical Dystonia; Transcranial direct current stimulation (tDCS); Transcranial magnetic stimulation (TMS); Sensorimotor network; Cerebellum; Non-invasive brain stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anodal ctDCS (Active Comparator): Patients receive anodal ctDCS stimulation for 20 minutes with 2 mA
  Interventions: Device: Anodal and cathodal ctDCS
- Cathodal ctDCS (Active Comparator): Patients receive cathodal ctDCS stimulation for 20 minutes with 2 mA
  Interventions: Device: Anodal and cathodal ctDCS
- Sham stimulation (Sham Comparator): Patients receive ctDCS stimulation for 20 minutes with 0 mA
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Anodal and cathodal ctDCS — CtDCS will be delivered using an DC-stimulator and two saline-soaked sponge electrodes: one electrode placed 3 cm lateral to the right of the inion, the other electrode on the right buccinator muscle. A 2 mA current will be delivered through these electrodes for a duration of 20 minutes with a 8-second fade-in and fade-out.
  Arms: Anodal ctDCS; Cathodal ctDCS
Device: Sham stimulation — The tDCS procedure will be identical to the active (anodal and cathodal) stimulation condition, but stimulation will cease after 30 seconds.
  Arms: Sham stimulation

SUMMARY:
Cervical dystonia (CD) is a movement disorder characterized by involuntary muscle contractions of the neck, leading to abnormal head postures and movement, pain and impaired motor function. Current treatments for CD, such as botulinum toxin injections and physical therapy, may not always provide sufficient relief of symptoms and may fail to offer long-term benefits for patients. As a result, new therapeutic approaches are needed. Transcranial direct current stimulation (tDCS) is a non-invasive brain stimulation technique that modulates neuronal activity. Recent neurophysiological studies suggest that cerebellar tDCS (ctDCS), in particular, could be beneficial in modulating the activity of the sensorimotor network in CD. This clinical trial aims to investigate the effects of ctDCS on the excitability of the sensorimotor network and motor symptom severity in CD patients. Applying transcranial magnetic stimulation (TMS) we will evaluate the effects of anodal, cathodal and sham ctDCS to improve the understanding of the neurophysiological mechanisms underlying CD and the potential therapeutic role of ctDCS.

DETAILED DESCRIPTION:
Dystonia is a movement disorder characterized by involuntary, sustained or intermittent muscle contractions, resulting in abnormal movements and postures. CD is the most common form of focal dystonia. It is characterized by abnormal postures or movements of the head. Standard treatment in patients with CD includes regular botulinum toxin injections and physical therapy, but many patients continue to experience symptoms, especially towards the end of the treatment cycle, highlighting the need for alternative treatment options.

One of the challenges in treating CD is the incomplete understanding of its underlying neurophysiological mechanisms. Recently, CD has been recognized as a network disorder, affecting the basal ganglia, the brainstem, the sensorimotor cortex and the cerebellum. So far, there is increasing evidence supporting the role of the cerebellum in the pathophysiology of dystonia, including animal models, neuroimaging and neurophysiological studies, but the exact the role in the proposed dystonia network is only incompletely understood.

TDCS is a form of non-invasive brain stimulation modulating the excitability of superficially located neurons. CtDCS is known to modulate the excitability of neurons of the cerebellar cortex, while the cerebellar nuclei and the brain stem remain unaffected. It has been shown that anodal ctDCS increases and cathodal ctDCS decreases the excitability of the cerebellum.

This randomized and sham-controlled clinical trial aims to investigate the effects of anodal and cathodal ctDCS in CD patients, focusing on both the sensorimotor network excitability and motor symptom severity. Participants will undergo three separated experimental sessions separated by one week, each with a different stimulation condition: anodal, cathodal, and sham ctDCS. Both, the study participants and the experimenter will be blinded to the order of stimulation mode.

The outcome measures will include:

1. Changes in the sensorimotor network before and after ctDCS stimulation, assessed by TMS. Measurements include four main metrics to determine the neurophysiological properties of the sensorimotor network in different ways:

   1. Single-pulse TMS (SP-TMS) of the left primary motor cortex, used to quantify the amplitude of motor-evoked potentials (MEPs) in response to unconditioned stimuli,
   2. Short-interval intracortical inhibition (SICI),
   3. Short-latency afferent inhibition (SAI),
   4. Cerebellar brain inhibition (CBI).
2. Clinical motor symptom severity, assessed with the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) before and after each session.

This study aims to improve the understanding of the neurophysiological mechanisms and clinical effects of ctDCS in isolated CD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of isolated cervical dystonia
* Written informed consent by the patient

Exclusion Criteria:

* History of other neurological disorders other than CD
* Secondary dystonia
* Severe head tremor
* Intake of centrally acting medication
* Contraindications to TMS, such as metallic implants, pregnancy and history of seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in sensorimotor network | Baseline (pre-intervention) and immediately after the intervention
  Before and after each tDCS intervention, TMS will be used to assess the neurophysiological properties of the sensorimotor network with four main metrics:
  1. Single-pulse TMS (SP-TMS):
     MEPs will be recorded from the right FDI in response to single-pulse TMS applied over the left primary motor cortex.
  2. Short-interval intracortical inhibition (SICI):
     SICI will be assessed using a paired-pulse TMS protocol, in which two stimuli are delivered at a short interstimulus interval over the primary motor cortex.
  3. Short-latency afferent inhibition (SAI):
     SAI consists of electrical conditioning stimuli to the right index finger preceding the test stimulus delivered by TMS to the left primary motor cortex.
  4. Cerebellar-brain-inhibition (CBI):
  To assess CBI, a conditioning stimulus will be applied over the right cerebellar hemisphere using a second magnetic coil, followed by a cortical test stimulus over the left primary motor cortex.

SECONDARY OUTCOMES:
Clinical symptom severity | Baseline (pre-intervention) and immediately after the intervention
  Each session will begin and end with a clinical evaluation using the TWSTRS to quantify motor symptom severity, disability and pain associated with CD.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ugawa Y, Uesaka Y, Terao Y, Hanajima R, Kanazawa I. Magnetic stimulation over the cerebellum in humans. Ann Neurol. 1995 Jun;37(6):703-13. doi: 10.1002/ana.410370603. PMID 7778843
- [Background] Porcacchia P, Alvarez de Toledo P, Rodriguez-Baena A, Martin-Rodriguez JF, Palomar FJ, Vargas-Gonzalez L, Jesus S, Koch G, Mir P. Abnormal cerebellar connectivity and plasticity in isolated cervical dystonia. PLoS One. 2019 Jan 25;14(1):e0211367. doi: 10.1371/journal.pone.0211367. eCollection 2019. PMID 30682155
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Background] Hamada M, Strigaro G, Murase N, Sadnicka A, Galea JM, Edwards MJ, Rothwell JC. Cerebellar modulation of human associative plasticity. J Physiol. 2012 May 15;590(10):2365-74. doi: 10.1113/jphysiol.2012.230540. Epub 2012 Apr 2. PMID 22473780
- [Background] Grimm K, Prilop L, Schon G, Gelderblom M, Misselhorn J, Gerloff C, Zittel S. Cerebellar Modulation of Sensorimotor Associative Plasticity Is Impaired in Cervical Dystonia. Mov Disord. 2023 Nov;38(11):2084-2093. doi: 10.1002/mds.29586. Epub 2023 Aug 28. PMID 37641392
- [Background] Brighina F, Romano M, Giglia G, Saia V, Puma A, Giglia F, Fierro B. Effects of cerebellar TMS on motor cortex of patients with focal dystonia: a preliminary report. Exp Brain Res. 2009 Feb;192(4):651-6. doi: 10.1007/s00221-008-1572-9. Epub 2008 Sep 25. PMID 18815775
- [Background] Albanese A, Bhatia K, Bressman SB, Delong MR, Fahn S, Fung VS, Hallett M, Jankovic J, Jinnah HA, Klein C, Lang AE, Mink JW, Teller JK. Phenomenology and classification of dystonia: a consensus update. Mov Disord. 2013 Jun 15;28(7):863-73. doi: 10.1002/mds.25475. Epub 2013 May 6. PMID 23649720